CLINICAL TRIAL: NCT05521594
Title: Accuracy of FNAC in Thyroid Nodules Compared to to Surgical Specimen : QOC Experience
Acronym: Thyroid FNAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qena Oncology Center (Other Government)
Responsible Party: Principal Investigator, Mohamed Ahmed Orabi, specialist of surgical oncology at Qena Oncology Center, Qena Oncology Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Qena Oncology Center 2
Record Dates: First submitted 2022-08-20; First posted 2022-08-30 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Fine Needle Aspiration Cytology; Thyroid Diseases
Keywords: FNAC; thyroid nodules; thyroidectomy
MeSH Terms: conditions — Thyroid Diseases; Thyroid Nodule

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FNAC (Experimental)
  Interventions: Procedure: Fine Needle Aspiration Cytology
- post operative hitopathology (Experimental)
  Interventions: Procedure: Fine Needle Aspiration Cytology

INTERVENTIONS:
Procedure: Fine Needle Aspiration Cytology — Comparison between FNAC and post operative specimen after thyroid surgery
  Other Names: Thyrodectomy

SUMMARY:
Thyroid gland diseases are the second most common endocrine disease following diabetes mellitus(1). Thyroid nodules are common disorders with a prevalence ranged from 4 to 7% in adult population, 5%-30% are malignant [1].Fine-needle aspiration cytology (FNAC) is an easy, cost-effective test for cancer diagnosis, and its use has markedly decreased the number of unnecessary thyroid surgeries(2).

DETAILED DESCRIPTION:
it should be noted that FNAC cannot differentiate between benign and malignant follicular neoplasms.differentiation between follicular adenoma and follicular carcinoma is only possible after thyroid lobectomy.[2,3] In addition, a study of FNAC showed that 68% of the cases diagnosed by FNAC as follicular neoplasm turned out to be the follicular type of papillary carcinoma, indicting a considerable overlap between benign and malignant neoplasms.[4] Incidental findings of thyroid nodules have increased exponen¬tially in recent years, mostly due to the widespread application of high-resolution ultrasound (US) to the thyroid [5].Several in¬ternational scientific societies have established clinic-radiolog¬ical guidelines for the diagnosis and the management of thy¬roid nodules [2,3]. The American College of Radiology identifies 5 radiological risk levels and recommends US-guided fine-nee¬dle aspiration cytology (US-FNAC) of high-suspicion nodules if 10 mm or larger, and of nodules with a low risk for malignan¬cy only if larger than 25 mm [2]. According to the European Thyroid Association Guidelines (EU-TIRADS), nodules with no high-risk features (oval-shaped, isoechoic/hyperechoic with smooth margins) should be considered at low risk and FNA performed only if greater than 20 mm, while high-risk nodules greater than 10 mm should undergo FNAC, with possible FNAC also in 5-10 mm nodules if highly suspicious [3].

ELIGIBILITY:
Inclusion Criteria:

* Thyroid diseases
* Multi nodullar
* single nodules
* diffuse goiter
* Thyroid diseases underwent FNAC Then Thyroid surgery

Exclusion Criteria:

* Patients with no diagnostic FNAC

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Incidence of true positive results of FNAC after thyroidectomy | 10 days
  Accuracy of FNAC in thyroid nodules compared to to surgical specimen : QOC experience
Percentage of malignant thyroid nodules not observed by FNAC | 10 days
  type of thyroid malignancy not observed by FNAC
Incidence of false negative results by FNAC | 10 days
  false negative that diagnosed by FNAC not malignant but proved malignancy after surgical excion
Percentage of Total number of true results of FNAC to the total number of cases | 10 days
  accuracy of FNAC

CONTACTS AND LOCATIONS:
Overall Officials: Amr M Makky, specialist surgical onclogy, Study Director — Qena Oncology Center- Medical Military Academy; Abdullah Atyah Ali, Ass.Lecture General Surgery, Study Director — Qena Oncology Center--Luxor University; Mohamed Ahmed Orabi, specialist surgical onclogy, Principal Investigator — Qena Oncology Center; Mina Romany Tawfeek, Study Chair — Qena Oncology Center; Mahmoud Ahmed Dosoky, specialist pathology, Study Director — Qena Oncology Center
Locations (1):
- Qena Oncology Center, Qina, Egypt

IPD SHARING:
Plan to Share IPD: Undecided